CLINICAL TRIAL: NCT01230255
Title: Percutaneous Catheter Decompression in the Treatment of Elevated Intra-abdominal Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orlando Regional Medical Center (Other)
Responsible Party: Michael L. Cheatham, MD, Orlando Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OH09.068.04
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Compartment Syndromes
Keywords: intra-abdominal pressure; intra-abdominal hypertension; abdominal compartment syndrome; open abdomen; percutaneous
MeSH Terms: conditions — Compartment Syndromes; Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous catheter decompression (Experimental): Ultrasound guided percutaneous catheter drainage of free intra-peritoneal fluid or blood
  Interventions: Procedure: Percutaneous catheter drainage
- Open abdominal decompression (Active Comparator): Surgical treatment of elevated intra-abdominal pressure through traditional open abdominal decompression
  Interventions: Procedure: Percutaneous catheter drainage

INTERVENTIONS:
Procedure: Percutaneous catheter drainage — Ultrasound guided insertion of a 14 French pigtail catheter to drain free intra-peritoneal fluid or blood and thereby reduce elevated intra-abdominal pressure

SUMMARY:
Intra-abdominal hypertension (IAH) and abdominal compartment syndrome (ACS) have traditionally been treated surgically through emergent laparotomy. Intensivist-performed bedside drainage of free intra-peritoneal fluid or blood [percutaneous catheter decompression (PCD)] has been suggested as a less-invasive alternative to traditional open abdominal decompression (OAD). This study assesses the relative efficacy of PCD vs. OAD in reducing elevated intra-abdominal pressure (IAP).

DETAILED DESCRIPTION:
Intra-abdominal hypertension (IAH), the presence of elevated intra-abdominal pressure (IAP), and abdominal compartment syndrome (ACS), the development of IAH-induced organ-dysfunction and failure, are both associated with significant morbidity and mortality when appropriate and expedient treatment is not rendered. Elevated IAP is an independent predictor of mortality during critical illness and serial IAP measurements are increasingly being performed in the intensive care unit (ICU) setting.

Despite growing evidence demonstrating the survival benefit of serial IAP monitoring and abdominal decompression in patients with IAH / ACS, some physicians are reluctant to consider decompression or unable to convince a surgeon to open the abdomen of patients manifesting IAH-related organ failure. Percutaneous catheter drainage (PCD) of free intra-abdominal fluid, air, abscess, or blood has been suggested in several case reports and small clinical trials to be a less invasive technique for reducing IAP and potentially correcting IAH-induced organ dysfunction. PCD, performed under ultrasound or computed tomography guidance, is described in the current World Society of the Abdominal Compartment Syndrome (WSACS) consensus recommendations as a therapeutic option, but insufficient data currently exist to support a strong evidence-based recommendation for the percutaneous treatment of IAH / ACS (10,12). Since 2007, we have employed PCD in the treatment of patients with IAH due to free intraperitoneal fluid and blood. This study describes our experience with the less invasive PCD technique compared to contemporaneous matched control patients who received traditional open abdominal decompression (OAD) for the treatment of IAH / ACS.

ELIGIBILITY:
Inclusion Criteria:

* Elevated intra-abdominal pressure

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction in intra-abdominal pressure | 4 hours

SECONDARY OUTCOMES:
Increased abdominal perfusion pressure | 4 hours
Percutaneous drainage failure rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Cheatham, MD, Principal Investigator — Orlando Regional Medical Center
Locations (1):
- Orlando Regional Medical Center, Orlando, Florida, United States